CLINICAL TRIAL: NCT02307045
Title: Effect of Smoking Reduction on Endothelial Glucocalyx and Arterial Wall Properites During Medically-aided Smoking Cessation Program.
Brief Title: Effect of Smoking Reduction on Endothelial Glucocalyx and Vascular Function
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Assistant Professor in Cardiology, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SMOKING-VAR-NIC-ATTIKON
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Smoking Cessation
Keywords: Arterial stiffness; Endothelial Glycocalyx
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline; Nicotine; Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- varenicline (Active Comparator): Stimulation of nicotinic receptors by varenicline (Champix) 1,0 mg po
  Interventions: Drug: Varenicline
- nicotine (Active Comparator): Nicotine replacement therapy with transdermal patches and/or chewing gums
  Interventions: Drug: nicotine

INTERVENTIONS:
Drug: Varenicline — Stimulation of nicotinic receptors by varenicline (Champix) 1,0 mg po
  Other Names: Champix (varenicline)
  Arms: varenicline
Drug: nicotine — Nicotine replacement therapy with transdermal patches and/or chewing gums
  Other Names: Nicorette (nicotine)
  Arms: nicotine

SUMMARY:
The integrity of endothelial glucocalyx plays a vital role in vascular permeability and inflammation. Smoking cessation is related with improved vascular function and is a key component of secondary cardiovascular prevention. Pharmacotherapy is a standard component of evidence based smoking cessation treatment. This study was designed to determine the effects medically-aided smoking cessation on glucocalyx thickness and arterial elasticity smoking cessation programs

DETAILED DESCRIPTION:
The investigators will examine smokers without cardiovascular disease treated with transdermal nicotine patches and/or varenicline at before, 4, 12, 24 and 48 weeks after treatment during validated smoking cessation program. The investigators will measure changes between baseline and 4,12,24, and 48 weeks after treatment of :

1. exhaled carbon monoxide (CO, ppm) and self-reported number of cigarretes/day
2. carotid-femoral pulse wave velocity (PWVc m/sec-Complior SP ALAM) and augmentation index (AI %-Arteriograph,TensioMed)
3. perfused boundary region (PBR) of the sublingual arterial microvessels (ranged from 5-25 micrometers) using Sideview Darkfield imaging (Microscan, Glycocheck). The PBR in microvessels is the cell-poor layer which results from the phase separation between the flowing red blood cells (RBC) and plasma. The PBR includes the most luminal part of glycocalyx that does allow cell penetration. Increased PBR is considered an accurate index of reduced endothelial glucocalyx thickness because of a for deeper penetration of the RBC in the glucocalyx
4. oxidative stress, thrombosis and inflammatory biomarkers in blood samples.

Non smokers of similar age and sex will serve as controls.

ELIGIBILITY:
Inclusion Criteria:

* Smokers

Exclusion Criteria:

* Coronary artery disease
* Heart failure
* Diabetes mellitus
* Dyslipidemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2014-12-03 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Changes in endothelial function between baseline and during medically-aided smoking cessation program. | Baseline, 1 month, 3 months, 6 months and 12 months.
  Changes in endothelial function between baseline and during medically-aided smoking cessation program as assessed by endothelial glycocalyx thickness.

SECONDARY OUTCOMES:
Changes in a composite of markers of vascular function between baseline and during medically-aided smoking cessation program. | Baseline, 1 month, 3 months, 6 months and 12 months.
  Changes in vascular function between baseline and during medically-aided as assessed by a composite of pulse wave velocity, augmentation index and central aortic blood pressure.
Follow up for cardiovascular events | baseline , ten years
  Association of endothelial glycocalyx as assessed by perfused boundary region (μm) with adverse cardiac events (composite of death, myocardial infarction, stroke , hospitalization for heart failure) during ten year follow -up in smokers and non-smoker subjects

CONTACTS AND LOCATIONS:
Overall Officials: Ignatios Ikonomidis, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; Kalliroi Kourea, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; George Pavlidis, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; Margarita Marinou, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; John Lekakis, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece
Locations (1):
- ''Attikon'' University General Hospital, Athens, Attica, Greece

REFERENCES:
- [Derived] Ikonomidis I, Marinou M, Vlastos D, Kourea K, Andreadou I, Liarakos N, Triantafyllidi H, Pavlidis G, Tsougos E, Parissis J, Lekakis J. Effects of varenicline and nicotine replacement therapy on arterial elasticity, endothelial glycocalyx and oxidative stress during a 3-month smoking cessation program. Atherosclerosis. 2017 Jul;262:123-130. doi: 10.1016/j.atherosclerosis.2017.05.012. Epub 2017 May 13. PMID 28549278